CLINICAL TRIAL: NCT00563745
Title: Randomised Trial on Telemedicine to Save Health Care Requests for Patients With Severe Chronic Respiratory Failure.
Brief Title: Telemedicine for Patients With Chronic Respiratory Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Vitacca (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Sponsor-Investigator, Michele Vitacca, Fondazione Salvatore Maugeri, Fondazione Salvatore Maugeri
Organization: Fondazione Salvatore Maugeri (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N°158
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Respiratory Failure
Keywords: COPD; ALS; Telemedicine; mechanical ventilation; Integrated care; strict follow up; impact and costs on health care resources; telemedicine programme; home mechanical ventilation (HMV); frail patients; chronic respiratory failure (CRF)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Experimental): Patients were submitted to a Telemedicine program for 1 year
  Interventions: Device: telemedicine program
- Control group (No Intervention): Patients were submitted to usual care (i.e: educational plan and outpatient visits every 3 months)

INTERVENTIONS:
Device: telemedicine program — One year TM with continuous (h 24) on call accessibility to a nurse and/or a pulmonologist, a web-based call centre and a pulse oxymetry tracing will be provided.
  Other Names: home care
  Arms: Telemedicine

SUMMARY:
In unstable patients needing oxygen and/or home mechanical ventilation, a nurse-centred TM programme (supported by continuous availability of a call centre and a pulsed oxygen system) is cost/effective saving health care resources.

DETAILED DESCRIPTION:
Background: Integrated care and strict follow up have been recommended for frail patients with chronic respiratory failure (CRF) discharged at home.

Objectives: To evaluate impact and costs on health care resources of a telemedicine programme (TM) for severe patients discharged at home with oxygen and/or home mechanical ventilation (HMV) with a high risk of hospital readmission.

Design: Prospective randomised controlled trial. Setting: Respiratory Rehabilitation Unit S. Maugeri Foundation between May 2004 and March 2007.

Participants: 240 CRF patients will be randomised into an intervention group (TM) and a control Group, which received current usual care (educational plan, 3 months outpatient visits).

Interventions: one year TM with continuous (h 24) on call accessibility to a nurse and/or a pulmonologist, a web-based call centre and a pulse oxymetry tracing.

Main outcome measures: survival, admissions to emergency room (ER), hospitalisations, urgent general practitioner (GP) calls, home relapses; probability to remain free from the above events will be also compared among groups. TM and health Care System costs as customer satisfaction will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* CRF patients discharged from Respiratory Unit with home MV

Exclusion Criteria:

* Severe co morbid conditions, i.e. lung cancer or other advanced malignancies, and extremely severe neurological disorders (with impaired cognitive status, ability to understand medical instructions, dementia or severe psychiatric illness)
* Logistical limitations due to extremely poor social conditions, such as illiteracy or no telephone access at home
* Being admitted to a nursing home
* Lack of caregiver when ventilated invasively (i.e. tracheal cannula with sounds uncertain) to allow a contact between care team and family
* Refusal to give informed consent

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate impact and costs on health care resources of a telemedicine programme (TM) for severe patients discharged with oxygen and/or home mechanical ventilation (HMV) with high risk of hospital readmission. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Principal Investigator — Fondazione S. Maugeri IRCCS
Locations (1):
- Telemedicine Service, Fondazione S. Maugeri, IRCCS, Lumezzane, Brescia, Italy

REFERENCES:
- [Background] Casas A, Troosters T, Garcia-Aymerich J, Roca J, Hernandez C, Alonso A, del Pozo F, de Toledo P, Anto JM, Rodriguez-Roisin R, Decramer M; members of the CHRONIC Project. Integrated care prevents hospitalisations for exacerbations in COPD patients. Eur Respir J. 2006 Jul;28(1):123-30. doi: 10.1183/09031936.06.00063205. Epub 2006 Apr 12. PMID 16611656
- [Background] Adams SG, Smith PK, Allan PF, Anzueto A, Pugh JA, Cornell JE. Systematic review of the chronic care model in chronic obstructive pulmonary disease prevention and management. Arch Intern Med. 2007 Mar 26;167(6):551-61. doi: 10.1001/archinte.167.6.551. PMID 17389286
- [Result] Vitacca M, Bianchi L, Guerra A, Fracchia C, Spanevello A, Balbi B, Scalvini S. Tele-assistance in chronic respiratory failure patients: a randomised clinical trial. Eur Respir J. 2009 Feb;33(2):411-8. doi: 10.1183/09031936.00005608. Epub 2008 Sep 17. PMID 18799512
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- See also: istitutional web site — http://www.fsm.it
- See also: telemedicine site — http://www.telemed.org
- See also: european telemedicine site — http://www.ehtel.org